CLINICAL TRIAL: NCT06653140
Title: Research on the Monitoring, Pathogen Screening, and Diagnostic System for Unexplained and Newly Emerging Acute Hepatitis
Status: Not yet recruiting | Type: Observational
Sponsor: Minghui Li (Other Government)
Responsible Party: Sponsor-Investigator, Minghui Li, Professor, Beijing Municipal Administration of Hospitals
Organization: Beijing Municipal Administration of Hospitals (Other Government)
Other Study IDs: 2023YFC2306901
Record Dates: First submitted 2024-10-09; First posted 2024-10-22 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis of Unknown Aetiology
Keywords: Unexplained hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, feces, liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will collect blood and liver tissue samples of unexplained and newly emerging acute hepatitis through a monitoring system. After excluding infections of hepatitis A-E viruses using enzyme immunoassay, chemical, and photometric methods to detect infection markers, multiplex PCR technology will be employed to screen for related pathogens. The goal is to establish a sensitive, rapid, and accurate diagnostic system.

DETAILED DESCRIPTION:
Unexplained hepatitis refers to cases where patients exhibit acute hepatitis symptoms that are not caused by hepatitis A, B, C, D, or E viruses, also known as non-hepatotropic viral hepatitis. On March 31, 2022, the UK first reported five cases of severe acute hepatitis of unknown origin in children. Subsequently, suspected cases were reported in multiple countries worldwide. As of November 2022, 1,010 cases have been reported in 35 countries, primarily affecting children under five years old, with approximately 5% of cases requiring liver transplantation, indicating a high severity rate. Possible causes of unexplained hepatitis include infections by viruses other than hepatitis viruses and autoimmune reactions. Newly emerging acute hepatitis refers to outbreaks of hepatitis caused by newly discovered pathogens or other factors. Research has indicated that the etiology and pathogenesis of unexplained hepatitis in children are related to infections by human adenovirus, adeno-associated virus 2 (AAV2), and cytomegalovirus. European countries conducted adenovirus testing on 457 children, with a positivity rate of 51.6% (236 cases). Two studies in the UK found high levels of AAV2 in the blood and liver samples of some children through metagenomic sequencing and PCR testing, although the specific pathogenesis remains unclear. Unexplained hepatitis and newly emerging acute hepatitis can cause a significant disease burden. Reports and discoveries in China are relatively rare. To accurately understand the incidence and pathogenic mechanisms of unexplained and newly emerging acute hepatitis in China, it is crucial to conduct monitoring, pathogen screening, and diagnostic system research. This project aims to collect blood and liver tissue samples of unexplained and newly emerging acute hepatitis through a monitoring system. After excluding infections of hepatitis A-E viruses using enzyme immunoassay, chemical, and photometric methods to detect infection markers, multiplex PCR technology and other methods will be employed to establish a pathogen detection platform for unexplained hepatitis. This will involve nucleic acid testing for common non-hepatotropic viruses that cause liver damage and constructing a stable multiplex PCR reaction system to achieve rapid screening and diagnosis of clinical samples. Understanding the incidence and dynamic trends of unexplained and newly emerging acute hepatitis, and studying their etiology and influencing factors through pathogen screening and diagnostic research, will provide technical support for the prevention and control of these conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Exhibiting symptoms of acute hepatitis;
2. Medical history, signs, and auxiliary examinations suggest hepatitis, but the cause is unknown or it is non-hepatotropic viral hepatitis;
3. Newly discovered pathogen infection or hepatitis caused by factors other than currently known ones;
4. The subject voluntarily participates in this study and signs the informed consent form.

Exclusion Criteria:

1. Patients with a clear etiology and diagnosis of hepatitis;
2. Patients who refuse to cooperate with sampling and sign the informed consent form;
3. Those deemed unsuitable for participation in this study by the researchers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Based on the suspected acute hepatitis case samples collected nationwide and the newly discovered suspected cases of unexplained and newly emerging acute hepatitis from the monitoring systems of the research centers participating in this study from 2024 to 2026.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Forms of outcomes | three years
  Validation of the Diagnostic Performance of the Monitoring Network and Early Warning System for Unexplained and Newly Emerging Acute Hepatitis

OTHER OUTCOMES:
Forms of outcomes | three years
  Research Report on the Types, Genotypes, Gene Mutations, and Evolutionary Molecular Characteristics of Pathogens Causing Newly Emerging Acute Hepatitis

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sergi CM. Acute Hepatitis of Unknown Origin (AHUO)-The Puzzle Ahead. Diagnostics (Basel). 2022 May 12;12(5):1215. doi: 10.3390/diagnostics12051215. PMID 35626370